CLINICAL TRIAL: NCT04017585
Title: Double Blind Randomized Clinical Trial in Subjects With Irritable Bowel Syndrome for the Identification of Gluten Sensitivity
Brief Title: Identification of Gluten Sensitivity in Irritable Bowel Syndrome
Acronym: IBS-NCGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Michele Barone, Professor, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Policlinic Hospital 5, Bari
Record Dates: First submitted 2019-07-08; First posted 2019-07-12 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Non-celiac Gluten Sensitivity; Irritable Bowel Syndrome
Keywords: gluten free diet; FODMAPs; gastrointestinal symptoms
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Interventional study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with IBS treated with gluten (Active Comparator): patients receiving gluten
  Interventions: Dietary Supplement: diet containing gluten
- patients with IBS treated with placebo (Placebo Comparator): patients receiving placebo
  Interventions: Dietary Supplement: Diet containing placebo

INTERVENTIONS:
Dietary Supplement: diet containing gluten — gluten will be added for 7 days to the low FODMAP/gluten free diet diet. After 1 week of wash-out, patients will switch (cross-over) to placebo for another 7 days
  Arms: patients with IBS treated with gluten
Dietary Supplement: Diet containing placebo — Placebo will be added for 7 days to the low FODMAP/gluten free diet diet. After 1 week of wash-out, patients will switch (cross-over) to gluten for another 7 days
  Arms: patients with IBS treated with placebo

SUMMARY:
The aim of our study will be to establish in how many subjects with gastrointestinal symptoms and previous diagnosis of irritable bowel syndrome (IBS), the clinical picture is attributable to non celiac gluten sensitivity (NCGS) or fermentable oligosaccharides, disaccharides, monosaccharides and polyols (FODMAPs) intolerance. For this purpose, all subjects with IBS will take a low FODMAPs diet, which implies the absence of cereals and consequently of gluten, and those presenting symptom improvement during this dietary treatment, will be exposed to a double-blind gluten or placebo challenge, to make a diagnosis of NCGS.

DETAILED DESCRIPTION:
Study design:

For this study, patients with diagnosis of IBS performed by Rome IV criteria and followed as outpatients at the Clinical Nutrition Clinic of "Petrucciani" Nursing Home of Lecce (LE), Italy, will be enrolled.

At baseline, the enrolled subjects will follow a balanced normal-caloric low-FODMAP and gluten-free diet for a period of 4 weeks. At the end of the 4 weeks patients who did not experience an improvement in symptoms will be considered "non-responders" and discontinue the clinical trial. Only those subjects who had showed a significant improvement in symptoms, will be enrolled for the phase 2 of the study that includes a challenge with gluten or with placebo, as described by the Salerno criteria.

ELIGIBILITY:
Inclusion Criteria:

* a gluten-containing diet for at least six months before enrollment
* anti-transglutaminase antibodies (IgA and IgG) absence
* normal serum IgA levels
* prick and specific IgE tests for wheat allergy negative

Exclusion Criteria:

* celiac disease
* wheat allergy
* chronic intestinal inflammatory diseases
* psychiatric disorders
* major abdominal surgery (in particular intestinal resections)
* diabetes mellitus
* previous anaphylactic episodes
* gluten-free diet in the previous six months
* pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Identification of FODMAP intollerance in IBS subjects | 4 weeks
  To evaluate the FODMAP intolerance, the response to a low FODMAP diet will be assessed by a visual analogue scale (VAS) before and after the dietary challenge. The VAS scale consists in is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptoms, pain, subjective feeling of well-being/malaise) orientated from the left (worst) to the right (best) The patient is invited to indicate a position (a point) along the line.
Identification of NCGS in IBS subjects who responded to low FODMAPs diet | 3 weeks
  To evaluate the NCGS, the response to the gluten challenge will be assessed by a visual analogue scale (VAS) before and after the dietary challenge. The VAS scale consists in is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptoms, pain, subjective feeling of well-being/malaise) orientated from the left (worst) to the right (best) The patient is invited to indicate a position (a point) along the line.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Barone, Study Director — University of Bari
Locations (1):
- Michele Barone, Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Catassi C, Elli L, Bonaz B, Bouma G, Carroccio A, Castillejo G, Cellier C, Cristofori F, de Magistris L, Dolinsek J, Dieterich W, Francavilla R, Hadjivassiliou M, Holtmeier W, Korner U, Leffler DA, Lundin KE, Mazzarella G, Mulder CJ, Pellegrini N, Rostami K, Sanders D, Skodje GI, Schuppan D, Ullrich R, Volta U, Williams M, Zevallos VF, Zopf Y, Fasano A. Diagnosis of Non-Celiac Gluten Sensitivity (NCGS): The Salerno Experts' Criteria. Nutrients. 2015 Jun 18;7(6):4966-77. doi: 10.3390/nu7064966. PMID 26096570
- [Result] Catassi C, Alaedini A, Bojarski C, Bonaz B, Bouma G, Carroccio A, Castillejo G, De Magistris L, Dieterich W, Di Liberto D, Elli L, Fasano A, Hadjivassiliou M, Kurien M, Lionetti E, Mulder CJ, Rostami K, Sapone A, Scherf K, Schuppan D, Trott N, Volta U, Zevallos V, Zopf Y, Sanders DS. The Overlapping Area of Non-Celiac Gluten Sensitivity (NCGS) and Wheat-Sensitive Irritable Bowel Syndrome (IBS): An Update. Nutrients. 2017 Nov 21;9(11):1268. doi: 10.3390/nu9111268. PMID 29160841
- [Result] Van den Houte K, Carbone F, Pannemans J, Corsetti M, Fischler B, Piessevaux H, Tack J. Prevalence and impact of self-reported irritable bowel symptoms in the general population. United European Gastroenterol J. 2019 Mar;7(2):307-315. doi: 10.1177/2050640618821804. Epub 2018 Dec 22. PMID 31080615
- [Result] Jones AL. The Gluten-Free Diet: Fad or Necessity? Diabetes Spectr. 2017 May;30(2):118-123. doi: 10.2337/ds16-0022. No abstract available. PMID 28588378
- [Result] Calasso M, Francavilla R, Cristofori F, De Angelis M, Gobbetti M. New Protocol for Production of Reduced-Gluten Wheat Bread and Pasta and Clinical Effect in Patients with Irritable Bowel Syndrome: A randomised, Double-Blind, Cross-Over Study. Nutrients. 2018 Dec 2;10(12):1873. doi: 10.3390/nu10121873. PMID 30513824
- [Result] Junker Y, Zeissig S, Kim SJ, Barisani D, Wieser H, Leffler DA, Zevallos V, Libermann TA, Dillon S, Freitag TL, Kelly CP, Schuppan D. Wheat amylase trypsin inhibitors drive intestinal inflammation via activation of toll-like receptor 4. J Exp Med. 2012 Dec 17;209(13):2395-408. doi: 10.1084/jem.20102660. Epub 2012 Dec 3. PMID 23209313
- [Result] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Result] Drossman DA. Functional Gastrointestinal Disorders: History, Pathophysiology, Clinical Features and Rome IV. Gastroenterology. 2016 Feb 19:S0016-5085(16)00223-7. doi: 10.1053/j.gastro.2016.02.032. Online ahead of print. PMID 27144617
- [Derived] Barone M, Gemello E, Viggiani MT, Cristofori F, Renna C, Iannone A, Di Leo A, Francavilla R. Evaluation of Non-Celiac Gluten Sensitivity in Patients with Previous Diagnosis of Irritable Bowel Syndrome: A Randomized Double-Blind Placebo-Controlled Crossover Trial. Nutrients. 2020 Mar 6;12(3):705. doi: 10.3390/nu12030705. PMID 32155878